CLINICAL TRIAL: NCT04278040
Title: Safety, Tolerability and Efficacy of Ultra-low Doses of Alkylating Drug Melphalan Inhalations for the Treatment of Non-cystic Fibrosis Bronchiectasis
Brief Title: Inhalations of Ultra-low Doses of Melphalan for the Treatment of Non-cystic Fibrosis Bronchiectasis
Acronym: SEADIB1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, Pulmonology Scientific Research Institute (Other Government)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Kirill Zykov, Deputy director for Science and Innovations, Federal State Budgetary Institution, Pulmonology Scientific Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSRI02-18
Record Dates: First submitted 2020-02-07; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: bronchiectasis; treatment; inhalation; low doses; alkylating drugs
MeSH Terms: conditions — Bronchiectasis; Respiratory Aspiration | interventions — Melphalan

STUDY DESIGN:
Masking Description: The trial was open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-cystic fibrosis bronchiectasis (NCFB) patients (Experimental): Inhalations with Melphalan 0,1 mg dissolved in 2 ml sodium chloride (NaCl) 0,9% 1 per day for 5 consequent days
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — Inhalations with low doses of Melphalan for 5 consequent days
  Other Names: Alkeran

SUMMARY:
This non-randomised open-label prospective pilot study evaluates the safety and efficacy of inhalations of ultra-low doses of alkylating drug melphalan for the treatment of non-cystic fibrosis bronchiectasis. All patients will receive 0,1 mg of melphalan in 5 daily inhalations 1 time per day.

DETAILED DESCRIPTION:
It was previously shown that in ultra-low (more than 100 times lower than conventional therapeutic) doses inhalations of alkylating drug (melphalan) are effective in severe steroid-resistant bronchial asthma, a form of the disease often characterized by neutrophilic type of inflammation. The exacerbation frequency reduced after the treatment, steroid-sparing effect was shown, morphological signs of bronchial epithelial regeneration were revealed and quality of life of asthmatic patients, treated with ultra-low doses of melphalan, improved. In preclinical studies and studies with volunteers, it was found that inhalations of ultra-low doses of melphalan do not have cytotoxic properties, but have local and systemic anti-inflammatory effects and decrease the activation of lymphocytes due to blockade of heavy β-chain of the interleukin (IL)-2 surface receptor. In addition, in ultra-low concentrations, alkylating agents are able to disrupt the cell signalling through the receptor for tumor necrosis factor, thereby exerting a protective effect from the cytotoxic activity of tumor necrosis factor (TNF)-α, which leads to the anti-inflammatory response. It can be assumed that the inhalation use of ultra-low doses of melphalan can be effective in patients with bronchiectasis, as in a disease characterized by a neutrophilic type of inflammation, leading to the improvement of quality of life, increasing the time to the first exacerbation and decreasing of exacerbation frequency.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Established diagnosis witn CT scan of non-cystic fibrosis bronchiectasis more than 12 months before the screening visit.
* Sputum expectoration not less than 3 months per year during more than 2 consecutive years
* Willing of the patient for cooperation

Non-Inclusion Criteria:

* Pregnant and lactating women and all women who are physiologically capable of becoming pregnant, who do not agree to use one or more of the following effective methods of contraception: intrauterine device or intrauterine system; hormonal contraception (implantable and oral preparations, patches); barrier methods of contraception; male sterilization (with appropriate documentation after a vasectomy about the absence of sperm in the ejaculate).

Effective contraception is used throughout the study until the last visit. "True abstinence" is acceptable only if it corresponds to the patient's preferred and habitual way of life.

Postmenopausal women (physiological menopause is defined as "no menstruation for 12 consecutive months") and women who have undergone sterilization surgery (for example, tubal occlusion, hysterectomy or bilateral salpingectomy) can be included in the study.

* A history of cystic fibrosis.
* Any exacerbation of respiratory infection requiring the use of systemic corticosteroids and / or antibiotics or hospitalization, which developed after the signing of the informed consent form and before the randomization visit (day 1, start of treatment). The criterion should be specified during the randomization visit.
* The presence of hemoptysis at the time of inclusion in the study.
* The presence of diseases of the respiratory tract, in addition to bronchiectasis, which can affect the effectiveness of the study drug and patient safety. Such conditions may include, among others, active tuberculosis, lung cancer, sarcoidosis, chronic obstructive pulmonary disease (COPD) IV (GOLD, 2017), uncontrolled bronchial asthma with respiratory failure, high pulmonary hypertension (> 25 mm Hg), interstitial lung disease, etc.
* Patients with a clinical significant disease of the cardiovascular system (for example, unstable angina, chronic heart failure New York Heart Association (NYHA) III / IV, acute myocardial infarction (within 6 months before inhalation of 1 dose), etc.
* Atrial fibrillation patients.
* Clinical significant 12-lead ECG abnormalities that may affect patient safety. The corrected QT interval (QTc) interval on the electrocardiogram (ECG in 12 leads) is more than 450 ms for men and more than 470 ms for women on screening and randomization visits.
* A history of hypersensitivity to any of the substances used in the study.
* Clinically significant deviations of laboratory parameters, indicating a significant or unstable concomitant disease, which may affect the effectiveness of the study drug or patient safety.
* Hemostasis deviation within 1 month before the first inhalation of the study drug, including confirmed:

  * Hemoglobin <10 g / 100 ml;
  * White blood cell count <3.0 x 10*9 / L;
  * The absolute number of neutrophils ≤ 1.5 x 10*9 / L;
  * Platelet count <100 x 10*9 / L.
* Unstable concomitant disease, such as uncontrolled hyperthyroidism, uncontrolled diabetes or other endocrine diseases; significant impairment of liver and kidney function; uncontrolled gastrointestinal diseases (for example, active peptic ulcer); uncontrolled neurological diseases; uncontrolled hematological diseases; uncontrolled autoimmune diseases or other diseases that, according to the researcher, may affect the effectiveness of the study drug and patient safety.
* Alcohol and/or drugs abuse 12 months before screening visit.
* Failure to perform tests to evaluate external respiration function, perform research procedures, or adhere to the treatment schedule provided for in the study.
* Participation in another clinical trial in which the study drug was administered less than 8 weeks before the screening visit.

Exclusion criteria:

* Informed consent withdrawn by the patient.
* The patient doesn't follow the instructions of the research staff regarding the requirements of the research protocol.
* Unable to contact patient.
* The researcher believes that participation in the study is not in the interests of the patient and / or further participation in the study is unsafe for the patient's health.
* There is a violation of the criteria for inclusion and / or non-inclusion in the study.
* The patient has developed adverse event, which, according to the researcher, makes further participation in the study unsafe for the patient.
* The licensing authority or ethics committee, for any reason, decides to discontinue the entire study or close this research center.
* A female patient becomes pregnant, is planning a pregnancy, or is breastfeeding while participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of drug-related side effects. | 6 months from the first inhalation
  The evaluation of side-effects, typical for the conventional therapeutic doses of melphalan (cough, bronchospasm, pulmonary fibrosis, interstitial pneumonitis; anorexia, gastrointestinal bleeding, ulcers of the stomach and duodenum, stomatitis, nausea, vomiting, esophagitis, diarrhea; myelodepression (leukopenia, thrombocytopenia, anemia), hemolytic anemia, bleeding and hemorrhage, vasculitis, veno-occlusive lesions, asystole; impaired urination, hematuria, hyperuricemia, nephropathy, edema, proteinuria, ovarian hypofunction, amenorrhea, azoospermia; anaphylaxis, anaphylactic shock, Quincke's edema, urticaria, skin rash, itching; dysfunction of the central nervous system, pain (back, side pain), the development of infections, fever, chills, alopecia, an increase in the concentration of 5-hydroxyindoleacetic acid, necrosis of the perivascular space, a feeling of heat and / or tingling at the injection site)

SECONDARY OUTCOMES:
The changes of The St George's Respiratory Questionnaire (SGRQ) | Day1 - Day 177 (±7 days)
  The evaluation of changes in quality of life with the SGRQ questionnaire (50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction). Scores are calculated for three domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. Lower score means a better the quality of life. A minimum change in score of 4 units was established as clinically relevant.
The changes of The Quality of Life-Bronchiectasis (QOL-B) questionnaire | Day1 - Day 177 (±7 days)
  The Quality of Life-Bronchiectasis (QOL-B), a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis bronchiectasis, contains 37 items on 8 scales (Respiratory Symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden).The minimal important difference score for the Respiratory Symptoms scale is 8.0 points. Higher scores represent a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Zykov, Prof, Principal Investigator — Federal State Budgetary Institution, Pulmonology Scientific Research Institute
Locations (1):
- Kirill Zykov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110
- [Background] Pukhalsky AL, Shmarina GV. Stimulatory and protective effects of alkylating agents applied in ultra-low concentrations. Pharmacology. 2001;62(3):129-32. doi: 10.1159/000056084. PMID 11287812
- [Background] Shmarina G, Pukhalsky A, Alioshkin V, Sabelnikov A. Melphalan reduces the severity of experimental colitis in mice by blocking tumor necrosis factor-alpha signaling pathway. Ann N Y Acad Sci. 2007 Jan;1096:97-105. doi: 10.1196/annals.1397.075. PMID 17405921
- [Background] Pukhalsky A, Shmarina G, Alioshkin V, Sabelnikov A. Alkylating drugs applied in non-cytotoxic doses as a novel compounds targeting inflammatory signal pathway. Biochem Pharmacol. 2006 Nov 30;72(11):1432-8. doi: 10.1016/j.bcp.2006.03.008. Epub 2006 Mar 14. PMID 16620792
- [Background] Pukhal'skii AL, Shmarina GV, Zykov KA, Aleshkin VA. [Effect of steroid therapy on the clinical course of bronchial asthma]. Vestn Ross Akad Med Nauk. 2009;(6):3-9. Russian. PMID 19645099
- [Background] Martinez-Garcia MA, Maiz L, Olveira C, Giron RM, de la Rosa D, Blanco M, Canton R, Vendrell M, Polverino E, de Gracia J, Prados C. Spanish Guidelines on the Evaluation and Diagnosis of Bronchiectasis in Adults. Arch Bronconeumol (Engl Ed). 2018 Feb;54(2):79-87. doi: 10.1016/j.arbres.2017.07.015. Epub 2017 Nov 9. English, Spanish. PMID 29128130
- [Background] Sinitsyn EA., Zykov KA. Non-cystic Fibrosis Bronchiectasis: Actual Problem Review and Treatment Prospects. Journal of Clinical Practice.2018;9(4):55-64. doi: https://doi.org/10.17816/clinpract9455-64
- [Background] Chalmers JD, Chotirmall SH. Bronchiectasis: new therapies and new perspectives. Lancet Respir Med. 2018 Sep;6(9):715-726. doi: 10.1016/S2213-2600(18)30053-5. Epub 2018 Feb 23. PMID 29478908